CLINICAL TRIAL: NCT01092013
Title: Comparative Evaluation of Simulator Based and Traditional In-surgery Laparoscopic Camera Training's Efficiency in Novices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Franzeck M Florian, cand. med., University of Zurich, Faculty of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: StV 12-2008
Record Dates: First submitted 2010-03-15; First posted 2010-03-24 (Estimated); Last update posted 2010-08-04 (Estimated); Status verified 2010-08

CONDITIONS: Laparoscopy; Clinical Competence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Operating room training (Active Comparator)
  Interventions: Behavioral: Training at actual laparoscopic surgery; Behavioral: Technical instruction
- Skills lab training (Active Comparator)
  Interventions: Behavioral: Training on laparoscopic simulator in skills lab; Behavioral: Technical instruction

INTERVENTIONS:
Behavioral: Training on laparoscopic simulator in skills lab — Laparoscopic camera training in a skills lab following training protocol for a total of 6 hours during 3 weeks.
  Arms: Skills lab training
Behavioral: Training at actual laparoscopic surgery — Assisting at 6 laparoscopic surgeries navigating the camera during 3 weeks
  Arms: Operating room training
Behavioral: Technical instruction — Technical instruction on proper handling of an angled laparoscope before randomization for 1 hour

SUMMARY:
This prospective randomized study aims for determination whether focused simulator based laparoscopic camera training in novices can improve camera performance in an actual clinical situations in the same manner as traditional training in the OR does, especially considering efficient use of training time.

DETAILED DESCRIPTION:
Medical students in their final years without any significant experience in handling an angled laparoscopic camera participate in the study and perform a camera guidance test in surgery. The participants are then randomized in two groups to receive either a simulator based or traditional in theatre training during three weeks. The camera test will be repeated, while both tests are going to be recorded. Videos of 14 camera tests carried out by laparoscopic experts are taped as well.

ELIGIBILITY:
Inclusion Criteria:

* Medical students on a surgical clerkship rotation at the department of visceral and transplantation surgery of the university hospital of Zurich, Switzerland

Exclusion Criteria:

* Any experience in laparoscopic camera handling in the OR and/or simulator based laparoscopic training

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Progress of skills shown in test regarding target centring as assessed by rating scale | After 3 weeks of individual training
  Students are sent to the OR to do two camera assessment tests involving a standardized set of tasks they had to accomplish operation. They had to center and hold for 5 seconds the following positions/organs and had to maintain the correct horizontal alignment during camera movement: 1. Left abdominal wall, 2. Descending colon, 3. Right lobe of liver, 4. Sigmoid colon 5. Caecum 6. Pelvis 7. Trocar entry site in the upper left quadrant 8. Desc. Colon. This assessment was video-taped. A rating scale quantifying target centring was used.

SECONDARY OUTCOMES:
Total time effort spend for respective training time | During 3 weeks of individual training
  Total time effort for OR group was defined as time used from receiving pager call (to go to OR) to leaving OR.
  Time effort for Skillslab group was defined as total time spend in Skillslab.
Progress of time to completion of test | After 3 weeks of individual training
Progress of skills shown in test regarding horizon alignment as assessed by rating scale | After 3 weeks of individual training
  Students are sent to the OR to do two camera assessment tests involving a standardized set of tasks they had to accomplish operation. They had to center and hold for 5 seconds the following positions/organs and had to maintain the correct horizontal alignment during camera movement: 1. Left abdominal wall, 2. Descending colon, 3. Right lobe of liver, 4. Sigmoid colon 5. Caecum 6. Pelvis 7. Trocar entry site in the upper left quadrant 8. Desc. Colon. This assessment was video-taped. A rating scale quantifying horizon alignment was used.

CONTACTS AND LOCATIONS:
Overall Officials: Florian M Franzeck, cand. med., Principal Investigator — University of Zurich, Faculty of Medicine; Dieter Hahnloser, MD, Study Director — University Hospital of Zurich, Departement of Visceral and Transplantation Surgery
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Franzeck FM, Rosenthal R, Muller MK, Nocito A, Wittich F, Maurus C, Dindo D, Clavien PA, Hahnloser D. Prospective randomized controlled trial of simulator-based versus traditional in-surgery laparoscopic camera navigation training. Surg Endosc. 2012 Jan;26(1):235-41. doi: 10.1007/s00464-011-1860-5. Epub 2011 Aug 19. PMID 21853391